CLINICAL TRIAL: NCT05221645
Title: Pembrolizumab in Combination With R-ICE Chemotherapy in Relapsed/Refractory Diffuse Large B-cell Lymphoma
Acronym: P+R-ICE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHMCAN1402
Record Dates: First submitted 2021-10-14; First posted 2022-02-03 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — pembrolizumab; Rituximab; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Intervention Model Description: The study has two treatment arms to which participants will be randomised on a 3:1 basis to the experimental arm. The control arm (Arm A) will be R-ICE for 3 cycles followed by an autologous stem cell transplant (for patients in a CR or PR on the post treatment PET-CT scan). The experimental arm (Arm B) will consist of P+R-ICE for 3 cycles followed by an autologous stem cell transplant (for patients in a CR or PR on the post treatment PET-CT scan) and maintenance Pembrolizumab every 3 weeks for one year.
  All patients will be randomised at study entry and will be stratified by relapse within 12 months or > 12 months of first line therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm A (Active Comparator): Patients will receive three cycles of R-ICE. Each cycle is 21 days +/- 3 days Rituximab 375mg/m2 Ifosfamide 5,000mg/m2 Carboplatin AUC = 5 (max dose 800mg) Etoposide 100mg/m2
  All patients who are deemed to be in CR or PR on the post treatment PET-CT scan will undergo autologous stem cell transplant (ASCT) within 4 weeks of completing R-ICE treatment. BEAM (carmustine, etoposide, cytarabine and melphalan) conditioning will be employed according to institutional protocol.
  Interventions: Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide
- Experimental Arm B (Experimental): Pembrolizumab 200mg Rituximab 375mg/m2 Ifosfamide 5,000mg/m2 Carboplatin AUC = 5 (max dose 800mg) Etoposide 100mg/m2 Patients will receive up to 3 cycles of: P+R-ICE, where each cycle is 21 days long +/-_3 days.
  All patients who are deemed to be in CR or PR on the post treatment PET-CT scan will undergo autologous stem cell transplant (ASCT) within 4 weeks of completing P+R-ICE treatment. BEAM (carmustine, etoposide, cytarabine and melphalan) conditioning will be employed according to institutional protocol.
  These patients will then be offered maintenance pembrolizumab every 3 weeks for one year.
  Interventions: Drug: Pembrolizumab; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a potent humanized immunoglobulin G4 (IgG4) monoclonal antibody (mAb) with high specificity of binding to the programmed cell death 1 (PD 1) receptor, thus inhibiting its interaction with programmed cell death ligand 1 (PD-L1) and programmed cell death ligand 2 (PD-L2). Based on preclinical in vitro data, pembrolizumab has high affinity and potent receptor blocking activity for PD 1. Pembrolizumab has an acceptable preclinical safety profile and is in clinical development as an intravenous (IV) immunotherapy for advanced malignancies. Keytruda® (pembrolizumab) is indicated for the treatment of patients across a number of indications because of its mechanism of action to bind the PD-1 receptor on the T cell.
  Other Names: KEYTRUDA
  Arms: Experimental Arm B
Drug: Rituximab — Rituximab is a chimeric mouse/human monoclonal antibody that binds to CD20, on pre-B and mature B lymphocytes and eliminates these cells potentially via a number of different mechanisms. Anti-CD20 mAbs, like rituximab, are classified by their CD20-binding characteristics, ability to induce complement-dependent cytotoxicity (CDC), and immune effector cell effects.
  Other Names: MabThera
Drug: Ifosfamide — Ifosfamide, Carboplatin and Etoposide (ICE) is proven to be an effective regimen in the relapsed refractory NHL population. In a study of 163 transplant eligible patients with relapsed/refractory disease, 66.3% of patients obtained CR/PR after 3 cycles of ICE chemotherapy at two weekly intervals.
Drug: Carboplatin — Ifosfamide, Carboplatin and Etoposide (ICE) is proven to be an effective regimen in the relapsed refractory NHL population. In a study of 163 transplant eligible patients with relapsed/refractory disease, 66.3% of patients obtained CR/PR after 3 cycles of ICE chemotherapy at two weekly intervals.
Drug: Etoposide — Ifosfamide, Carboplatin and Etoposide (ICE) is proven to be an effective regimen in the relapsed refractory NHL population. In a study of 163 transplant eligible patients with relapsed/refractory disease, 66.3% of patients obtained CR/PR after 3 cycles of ICE chemotherapy at two weekly intervals.

SUMMARY:
This is an open-label, multicentre, randomised phase II trial in relapsed or refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
The study has two treatment arms to which participants will be randomised on a 3:1 basis to the experimental arm. The control arm (Arm A) will be R-ICE for 3 cycles followed by an autologous stem cell transplant (for patients in a CR or PR on the post treatment PET-CT scan). The experimental arm (Arm B) will consist of P+R-ICE for 3 cycles followed by an autologous stem cell transplant (for patients in a CR or PR on the post treatment PET-CT scan) and maintenance Pembrolizumab every 3 weeks for one year.

All patients will be randomised at study entry and will be stratified by relapse within 12 months or > 12 months of first line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CD20 +ve diffuse large B-cell lymphoma, preferably with sufficient diagnostic material, obtained either at diagnosis or relapse (the latter is preferable) that is available to forward to the Haematological Malignancies Diagnostic Service (HMDS) for gene expression profiling and central pathology review
* Refractory to, or relapsed following, first-line or second-line treatments with rituximab concurrently with anthracycline or anthracenedione-based chemotherapy or similar (etoposide allowed if comorbid).

Refractory disease must fulfil one of the following:

* Continuing partial response (PR) from termination of first-line treatment. It is strongly recommended the lymphoma be reconfirmed by biopsy however, if these procedures are deemed to be inappropriate, the CI may determine eligibility following review of the imaging results and disease history.
* Continuing stable disease (SD) from termination of first-line treatment. Reconfirmation of the lymphoma by biopsy (preferred) is recommended but not mandatory.
* Progressive disease (PD). Biopsy or reconfirmation of the lymphoma is recommended but not mandatory.

  * Potentially eligible for high-dose therapy and peripheral blood progenitor cell rescue in the event of response
  * Positive lesions shown on baseline PET-CT must be compatible with CT defined anatomical tumour sites.
  * At least 2 demarcated lesions/nodes with a long axis >1.5 cm and a short axis equal to 1.0cm or 1 clearly demarcated lesion/node with a long axis >2.0cm and short axis of 1.0cm
  * Previous therapy related toxicity should have resolved to a grade that the investigator deems appropriate to commence further treatment
  * ECOG Performance Status 0 - 1
  * Has provided written informed consent
  * Willing to use acceptable contraception (see Section 4.6)
  * Aged 18 or over

Exclusion Criteria:

* Previous lymphoma cancer treatment beyond third line
* Radiotherapy or cytotoxic drugs within two weeks of trial treatment
* Major surgery within 4 weeks of trial registration. If a subject had major surgery, more than 4 weeks ago, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
* Treatment with any unlicensed drug within 4 weeks of trial treatment
* History of stroke or intracranial haemorrhage within 6 months prior to registration
* Pre-existing peripheral neuropathy grade >2
* Clinically significant cardiac disease (inc. unstable angina, acute myocardial infarction, congestive heart failure, a current LVEF of <40%) within 6 months of registration
* Any significant uncontrolled medical condition or known hypersensitivity to the study drugs
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis and tuberculosis.
* Other past or current malignancy within 2 years prior to registration unless in the opinion of the investigator it does not contraindicate participation in the study. Subjects who have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma, are eligible
* Known CNS involvement
* Serological positivity for Hepatitis B, C, or known HIV infection. As per standard of care, prior to initiation of immunochemotherapy, the results of hepatitis serology should be known prior to commencement of therapy.

Positive test results for chronic HBV infection (defined as positive HBsAg serology) will not be eligible.

Patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) will not be eligible.

Patients who have protective titres of hepatitis B surface antibody (HBsAb) after vaccination will be eligible.

Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA

* Screening laboratory values :

  * platelets <75x109/L (unless due to lymphoma involvement of the bone marrow)
  * neutrophils <1.0x109/L (unless due to lymphoma involvement of the bone marrow)
  * creatinine >2.0 times upper normal limit (unless due to lymphoma or unless creatinine clearance >50mL/min)
  * total bilirubin >1.5 times upper normal limit (unless due to lymphoma or a known history of Gilbert's disease)
  * ALT/AST >2.5 times upper normal limit (unless due to lymphoma)
  * alkaline phosphatase >2.5 times upper normal limit (unless due to lymphoma)
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis (Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone will be eligible as will be patients with controlled Type I diabetes mellitus on a stable dose of insulin).
* Patients who have previously undergone allogeneic transplantation.
* Live vaccination within 28 days of study treatment.
* Pregnant or lactating females. Women of child-bearing potential should have negative pregnancy test.
* History of severe allergic anaphylactic reactions to chimeric, human or humanised antibodies, or fusion proteins.
* History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Known hypersensitivity to CHO cell products or any component of the pembrolizumab formulation.
* Previous treatment with an anti-PD-1, anti-PD-L1 or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Corticosteroid use >10 mg/day of prednisolone or equivalent, for purposes other than for lymphoma symptom control.

Patients receiving corticosteroid treatment with <10 mg/day of prednisolone or equivalent must be documented to be on a stable dose of at least 4 weeks' duration prior to the start of Cycle 1. If glucocorticoid treatment is urgently required for lymphoma symptom control prior to the start of study treatment, prednisolone 100 mg or equivalent could be given for a maximum of 14 days as a pre-phase. A dose of up to 10mg or prednisolone or equivalent may be used during the screening phase to control symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish the event-free survival at 1 year in patients treated with P+R-ICE | 12 months
  Event free survival at 1 year (binary) - the proportion of patients alive and event free at 1 year. An event is defined as any of the following:
  * Progression / relapse of lymphoma
  * Stable disease at 3 cycles of therapy
  * Commencement of any unplanned non-protocol treatment for lymphoma
  * Death from any cause

SECONDARY OUTCOMES:
Event free survival (EFS) (time to event outcome) - median and at 1 and 2 years from Kaplan-meier curve | 12 months to 24 months
  Event free survival (EFS) (time to event outcome) - median and at 1 and 2 years from Kaplan-meier curve - defined as time from day of registration until relapse or progression, unplanned re-treatment of lymphoma, or death as a result of any cause, whichever occurs first. Patients who do not experience an EFS event will be censored at the date of their last clinical follow-up.
Progression-free survival (PFS) (time to event outcome) - median and at 1 and 2 years from Kaplan-meier curve | 12 months to 24 months
  Progression-free survival (PFS) (time to event outcome) - median and at 1 and 2 years from Kaplan-meier curve - defined as the time from the day of registration to the date of progression or death from any cause, whichever occurs first. Patients who do not experience progression, or death will be censored at the date of their last clinical follow up.
Overall Survival (OS) (time to event outcome) - median and at 1 and 2 years from Kaplan-meier curve | 12 months to 24 months
  Overall Survival (OS) (time to event outcome) - median and at 1 and 2 years from Kaplan-meier curve - defined as the time from the day of registration to the date of death from any cause. Patients who do not die will be censored at the date of their last follow up.
Number of patients achieving 2 x 106 CD34 positive cells per kg stem cells on harvest | 12 months
  Number of patients achieving 2 x 106 CD34 positive cells per kg stem cells on harvest
The number and proportion of patients achieving CR at the end of induction | 12 months
  The number and proportion of patients achieving CR at the end of induction (assessed by PET-CT at the end of cycle 3) determined by the Lugano response criteria
The number and proportion of patients achieving CR at the end of transplantation. | 12 months
  The number and proportion of patients achieving CR at the end of transplantation (PET-CT at week 27) determined by the Lugano response criteria. The Lugano response criteria determines a patient's response to treatment using a 1-4 staging to describe the spread of disease. Stage 1 being minimum spread of disease to stage 4 which is classed as a wide spread into at least one organ outside the lymph system. Clinicians will determine the Lugano response stage via a PET-CT image.
Number and proportion of patients achieving CR at any point during follow up. | 12 months
  Number and proportion of patients achieving CR at any point during follow up determined by the Lugano response criteria. The Lugano response criteria determines a patient's response to treatment using a 1-4 staging to describe the spread of disease. Stage 1 being minimum spread of disease to stage 4 which is classed as a wide spread into at least one organ outside the lymph system. Clinicians will determine the Lugano response stage via a PET-CT image.
Number and proportion of patients with an Objective response at end of cycle 3. | 12 months
  Number and proportion of patients with an Objective response (partial or complete metabolic response (PR or CR)) at end of induction assessed by PET-CT at end of cycle 3 determined by the Lugano response criteria. The Lugano response criteria determines a patient's response to treatment using a 1-4 staging to describe the spread of disease. Stage 1 being minimum spread of disease to stage 4 which is classed as a widespread into at least one organ outside the lymph system. Clinicians will determine the Lugano response stage via a PET-CT image.
Number and proportion of patients with an Objective response at the end of transplantation. | 12 months
  Number and proportion of patients with an Objective response (partial or complete metabolic response (PR or CR)) assessed by PET-CT at the end of transplantation (week 27) as determined by the Lugano response criteria. The Lugano response criteria determines a patient's response to treatment using a 1-4 staging to describe the spread of disease. Stage 1 is the minimum spread of disease to stage 4 which is classed as a widespread into at least one organ outside the lymph system. Clinicians will determine the Lugano response stage via a PET-CT image.
Number and proportion of patients achieving an Objective response at any time point. | 12 months
  Number and proportion of patients achieving an Objective response (CR or PR) at any point during follow up determined by the Lugano response criteria. The Lugano response criteria determines a patient's response to treatment using a 1-4 staging to describe the spread of disease. Stage 1 being the minimum spread of disease to stage 4 which is classed as a widespread into at least one organ outside the lymph system. Clinicians will determine the Lugano response stage via a PET-CT image.
Frequency, severity and causality of adverse and serious adverse events. | 12 months
  Frequency, severity and causality of adverse and serious adverse events severity according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Oxford Cancer & Haematology Centre, The Churchill Hospital, Headington, Oxford
  - The Beatson West of Scotland Cancer Centre, Glasgow

IPD SHARING:
Plan to Share IPD: No